CLINICAL TRIAL: NCT03114267
Title: Involvement of Viral Infections in the Pathogenesis of Chronic Lymphocytic Thyroiditis
Acronym: Etude thyrovir
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI11-PR-DESAILLOUD-1
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Autoimmune Diseases; Chronic Lymphocytic Thyroiditis
MeSH Terms: conditions — Autoimmune Diseases; Hashimoto Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with chronic lymphocytic thyroiditis
  Interventions: Other: Comparison of the prevalences of the parvovirus genome
- Healthy subjects
  Interventions: Other: Comparison of the prevalences of the parvovirus genome

INTERVENTIONS:
Other: Comparison of the prevalences of the parvovirus genome — Comparison of the prevalences of the parvovirus genome between cases and controls and then of other viruses according to the results of parvoviruses and data from the literature

SUMMARY:
Autoimmune diseases represent a heterogeneous group of pathologies whose etiopathogenic mechanisms are most often unknown. Autoimmune diseases are the leading cause of morbidity and mortality in young women and autoimmune thyroid diseases are the most common.

Viral infections are the main environmental factors suspected of triggering autoimmune diseases. Several viruses are certainly involved, all of which are possibly capable of triggering an autoimmune response. However, the precise identification of the viruses involved remains to be established.

It has been shown for the first time by the 2005 PHRC that enteroviral RNA is present in perioperative specimens of thyroid tissue. However, this case-control study did not show any difference between the thyroid group and the group other thyroid pathologies It has been recently published that Parvovirus is possibly involved in thyroiditis: the parvoviral genome is present in the thyroid tissue of Hashimoto thyroiditis operated and more precisely is present within the thyrocytes itself.

ELIGIBILITY:
Inclusion Criteria:

* Patients participating in PHRC 2005 "involvement of enteroviruses in TLC pathogenesis"
* Inclusion of TLC: presence of a significant lymphocyte infiltrate within the thyroid parenchyma defined by the presence of clusters of more than 30 to 50 lymphocytes
* Inclusion of controls: absence of significant lymphocyte infiltrate

Exclusion Criteria:

* Persons refusing to participate in research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were recruited after PHRC 2005. Written information for the extension of the study will be sent with a copy of the summary of the scientific publication on Enterovirus (PHRC 2005).
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2012-01-06 (Actual); Primary Completion 2015-01-06 (Actual); Study Completion 2015-01-06 (Actual)

PRIMARY OUTCOMES:
Analysis of the viral genome by PCR carried out in the Virology department, Analysis of the presence of capsid protein | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France